CLINICAL TRIAL: NCT00640328
Title: A Double-blind, Randomized, Placebo Controlled, Multicenter, Dose-finding Trial of Ofatumumab in Relapsing Remitting Multiple Sclerosis (RRMS) Patients
Brief Title: Ofatumumab Dose-finding in Relapsing Remitting Multiple Sclerosis (RRMS) Patients
Acronym: OMS115102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115102; NCT01526993 (obsolete NCT alias)
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: relapsing forms of multiple sclerosis; ofatumumab; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1.1 (Experimental): 100mg ofatumumab then placebo
  Interventions: Drug: Ofatumumab 100; Drug: Placebo
- Cohort 1.2 (Experimental): placebo then 100mg ofatumumab
  Interventions: Drug: Ofatumumab 100; Drug: Placebo
- Cohort 2.1 (Experimental): 300mg ofatumumab then placebo
  Interventions: Drug: Ofatumumab 300; Drug: Placebo
- Cohort 2.2 (Experimental): placebo then 300mg ofatumumab
  Interventions: Drug: Ofatumumab 300; Drug: Placebo
- Cohort 3.1 (Experimental): 700mg ofatumumab then placebo
  Interventions: Drug: Ofatumumab 700; Drug: Placebo
- Cohort 3.2 (Experimental): placebo then 700mg ofatumumab
  Interventions: Drug: Ofatumumab 700; Drug: Placebo

INTERVENTIONS:
Drug: Ofatumumab 100 — 100mg
  Arms: Cohort 1.1; Cohort 1.2
Drug: Ofatumumab 300 — 300mg
  Arms: Cohort 2.1; Cohort 2.2
Drug: Ofatumumab 700 — 700mg
  Arms: Cohort 3.1; Cohort 3.2
Drug: Placebo — matching placebo

SUMMARY:
The trial consists of a dose escalation, to establish the safety of ofatumumab in RRMS patients. A 48-week treatment period followed by an individualized follow-up period until normalization of peripheral B-cell counts or Immunoglobulin G (IgG) levels.

DETAILED DESCRIPTION:
The trial consists of two phases, a 48 week treatment period, followed by an individualized treatment period of up to two years.

Patients are treated in cohorts of increasing doses (100 mg, 300 mg and 700 mg) with 12 patients in each dose cohort. Within each cohort patients are randomized asymmetrically in a 2:1 ratio such that eight patients will receive ofatumumab and four patients will receive placebo. After 24 weeks the patients randomized to placebo will be treated with the active dose for the cohort. For blinding purposes, patients randomized to the active dose will be treated with placebo after 24 weeks. Thus, each patient will receive two administrations of trial product with 24 weeks follow-up resulting in a total treatment period of 48 weeks duration. An Independent Data Monitoring Committee (IDMC) will review and evaluate the safety data of each cohort, a minimum of 4 weeks data including the week 4 Magnetic Resonance Imaging (MRI) from at least 10 patients, to consider if progression to the next higher dose cohort is acceptable.

The trial product is administered as two infusions separated by two weeks. Clinical assessment and Gadolinium enhanced (Gd-enhanced) MRI scan will be performed at weeks -4, 0, 2, 4, and every 4 weeks until week 48. The MRI scan at week 2 is carried out for safety assessment prior to administering the second infusion in the first treatment course. When patients in all dose cohorts have been dosed and have had week 4 MRI scans performed, an IDMC will review all available safety data.

After completion of week 48 patients will be followed to monitor B-cell and IgG normalization. B-cell levels will be monitored every 12 weeks until CD19+ cells have returned to baseline level (Visit 3) or normalized level. If the B-cell levels are not normalized after two years the patient should be followed until either the IgG or the B-cell levels are normalized (see Section 9.2.4 for details). During this period Gd-enhanced MRI follow up scans will be performed every 12 weeks to evaluate potential rebound, safety and for Progressive Multifocal Leukoencephalopathy (PML) monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with definite diagnosis of relapsing-remitting MS according to McDonald criteria
* Patients with:
* At least two confirmed relapses within the last 24 months or
* At least one confirmed relapse within the last 12 months or
* One confirmed relapse between 12 and 24 months prior to screening, and at least one documented T1 Gd-enhancing lesion on an MRI performed within 12 months prior to screening.
* Patients with disability equivalent to Expanded Disability Status Scale (EDSS) score of 0-5.0 (both included) at screening
* Neurologically stable patients with no evidence of relapse for at least 30 days prior to start of Screening and during the Screening Phase
* Female patients must be either post-menopausal, surgically incapable of bearing children or practicing an acceptable method of birth control e.g. hormonal contraceptives, intrauterine device, spermicide and barrier as long as they are on trial medication and for a period of 1 year following the last infusion of trial drug. Females of childbearing potential must have a negative pregnancy test at screening visit prior to entry into the treatment period
* Following receipt of verbal and written information about the trial, the patient must provide signed informed consent before any trial related activity is carried out.

Exclusion Criteria:

* Diagnosis of Secondary Progressive Multiple Sclerosis (SPMS), Primary Progressive Multiple Sclerosis (PPMS) or Progressive Relapsing Multiple Sclerosis (PRMS) or Neuromyelitis optica
* Neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML) or confirmed PML
* Findings on brain MRI scan indicating any other clinically significant brain abnormality other than MS
* Patients unable to undergo MRI scans (e.g. due to pacemaker, severe claustrophobia, hypersensitivity to contrast media) or who lack adequate peripheral venous access
* Patients who have had the following treatments:
* Lymphocyte-depleting therapies (e.g. alemtuzumab (Campath®), anti-Cluster of Differentiation (CD4), cladribine, total body irradiation, bone marrow transplantation), mitoxantrone or cyclophosphamide at any time
* Anti-CD20 treatments or any monoclonal antibodies at any time
* Immunoglobulin, azathioprine, cyclosporine, tacrolimus or other immunosuppressive agents, immunomodulatory agents or plasma exchange within six months prior to randomization in the trial apart from Glatiramer Acetate and Interferon Beta (IFN-b).
* Glatiramer Acetate or IFN-b within three months prior to the randomization in the trial.
* Glucocorticoids or Adrenocorticotropic Hormone (ACTH) within one month prior to the screening in the trial.
* Receipt of a live vaccine within one month prior to screening in the trial.
* Plasmapheresis for treatment of relapses within 2 months prior to randomization in the trial.
* Initiation of therapy with Statins or hormone replacement treatment within one month or less prior to screening in the trial.
* Patients who have received other disease modifying therapies for MS may be allowed on a case to case basis after discussion with the sponsors medical monitor
* Past or current history of medically significant adverse effects (including allergic reactions) from:
* Cetirizine
* Prednisolone
* Paracetamol/acetaminophen
* Plasma proteins or a known hypersensitivity to components of the investigational product.
* Past or current malignancy, except for
* Cervical carcinoma Stage 1B or less
* Non-invasive basal cell and squamous cell skin carcinoma
* Cancer diagnoses with a complete response of a duration of > 5 years. Patients with a prior history of hematological malignancies are excluded regardless of response
* Clinically significant cardiac disease, including acute myocardial infarction within six months from screening, unstable angina, congestive heart failure, previous venous or arterial thrombosis or arrhythmia requiring therapy.
* Electrocardiogram (ECG) showing significant abnormality that the treating investigator determines may jeopardize the subject's health (i.e. acute ischemia, left bundle branch or bifascicular block)
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, immunodeficiency syndrome, pulmonary, cerebral, psychiatric or neurological disease which may impair their reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
* History of severe, clinically significant Central Nervous System (CNS) trauma (e.g. cerebral contusion, spinal cord compression) or a history or presence of myelopathy due to spinal cord compression by disk or vertebral disease
* Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C. Any previous serious infections should be discussed with the sponsors medical monitor (e.g. opportunistic or atypical infections)
* Female patients who are pregnant or nursing.
* Use of an investigational drug or other experimental therapy for a condition other than MS within 4 weeks prior to screening. Any prior use of an investigational drug or other experimental therapy for MS at any time should be discussed with the medical monitor.
* Current participation in any other interventional clinical trial. Participation in non-interventional trial requires approval of the protocol by the sponsor
* Serum vitamin B12 below lower limit of normal
* Positive polymerase chain reaction (PCR) screening for John Cunningham Virus (JC Virus) as measured by qualitative plasma and/or white blood cell JCV DNA
* Serologic evidence of Hepatitis B (HB) infection based on the results of testing for Hepatitis B Surface Antigen (HBsAg), anti- Hepatitis B Core (HBc) and anti- Hepatitis B Surface (HBs) antibodies with eligibility based on the results as follows:
* Patients positive for HBsAg are excluded
* Patients negative for HBsAg but positive for both anti-HBc and anti-HBs antibodies (indicating past infection) are eligible
* Patients negative for HBsAg and anti-HBc antibody but positive for anti-HBs antibody (indicating past vaccination) are eligible
* Patients negative for HBsAg and anti-HBs antibody but positive for anti-HBc antibody will require clarification of their status by testing for HB DNA, which if positive will exclude the patient from participation
* Patient with documented vaccination against Hepatitis B (primary and secondary immunization and booster) will be considered eligible for the trial.
* Positive serology for HIV
* Screening laboratory values:
* White Blood Cell (WBC) < 3.0 x 109/L
* Neutrophils < 2 x 109/L
* Platelets < 100 x 109/L
* Circulating IgG level < lower limit of normal (according to central laboratory range)
* Serum Alanine Aminotransferase (S-ALAT) > 2.5 times the upper limit of normal (according to central laboratory range)
* Serum Alpha Fetoprotein (S-AP) > 2.0 times the upper limit of normal (according to central laboratory range)
* Serum Aspartate Aminotransferase (ASAT) >3.0 times the upper limit of normal (according to central laboratory range)
* Bilirubin > 1.5 times the upper limit of normal (according to central laboratory range)
* S-creatinine > the upper limit of normal (according to central laboratory range)
* CD4 count <500 cells/mm3, CD4:CD8 <0.9
* Patients known or suspected of not being able to comply with a trial protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
* Positive test for Hepatitis C antibody confirmed with a Hepatitis C real time (RT) PCR assay.

Patients who are positive for Hepatitis C antibody and negative when the Hepatitis C RT PCR assay is performed will be eligible for the study. Patients who are positive for Hepatitis C antibody and have a positive or indeterminate result when the Hepatitis C RT PCR assay is performed will not be eligible for the study.

* Positive test results for tuberculosis using the QuantiFERON test and/or Chest X-ray findings suggestive of tuberculosis (TB). For patients who have had a Chest X-ray performed within the past 6 months without any findings indicative of TB, QuantiFERON test alone may be performed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In all 3 dose cohorts, participants in the active/placebo group received treatment with ofatumumab during the First Treatment Period and placebo during the Second Treatment Period. Participants in the placebo/active group received treatment with placebo during the First Treatment Period and ofatumumab during the second treatment period.
Groups:
- 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo: Ofa was administered as two doses of 100 mg via intravenous (iv) infusions separated by 2 weeks (wks) during the first 24-wk treatment period. Matching placebo was administered as two iv infusions separated by 2 wks during the second 24-wk treatment period. An Independent Data Monitoring Committee (IDMC) evaluated the safety data at Week 4 for participants receiving the 100 mg dose before considering progression to the 300 mg dose. After completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.
- 300 mg Ofa/Matching Placebo: Ofa was administered as two doses of 300 mg via iv infusions separated by 2 wks during the first 24-wk treatment period. Matching placebo was administered as two iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 300 mg dose before considering progression to the 700 mg dose. After completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.
- 700 mg Ofa/Matching Placebo: Ofa was administered as two doses of 700 mg via iv infusions separated by 2 wks during the first 24-wk treatment period. Matching placebo was administered as two iv infusions separated by 2 wks during the second 24-wk treatment period. After completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.
- Matching Placebo/100 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 100 mg via iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 100 mg dose before considering progression to the 300 mg dose. After completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.
- Matching Placebo/300 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 300 mg via iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 300 mg dose before considering progression to the 700 mg dose. After completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.
- Matching Placebo/700 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 700 mg via iv infusions separated by 2 wks during the second 24-wk treatment period. After completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.
Period: First Treatment Period (Weeks 0-24)
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Started | 8 | 11 | 7 | 4 | 4 | 4
Completed | 8 | 10 | 7 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Second Treatment Period (Weeks 24-48)
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Started | 8 | 10 | 7 | 4 | 4 | 4
Completed | 8 | 10 | 7 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: IFUP (Week 48 to Individual Termination)
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Started | 8 | 11 | 7 | 4 | 4 | 4
Completed | 8 | 10 | 6 | 3 | 4 | 4
Not Completed | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Not Recommended - Informed Consent Form | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo: Ofa was administered as two doses of 100 mg via intravenous (iv) infusions separated by 2 weeks (wks) during the first 24-wk treatment period. Matching placebo was administered as two iv infusions separated by 2 wks during the second 24-wk treatment period. An Independent Data Monitoring Committee (IDMC) evaluated the safety data at Week 4 for participants receiving the 100 mg dose before considering progression to the 300 mg dose.
- 300 mg Ofa/Matching Placebo: Ofa was administered as two doses of 300 mg via iv infusions separated by 2 wks during the first 24-wk treatment period. Matching placebo was administered as two iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 300 mg dose before considering progression to the 700 mg dose.
- 700 mg Ofa/Matching Placebo: Ofa was administered as two doses of 700 mg via iv infusions separated by 2 wks during the first 24-wk treatment period. Matching placebo was administered as two iv infusions separated by 2 wks during the second 24-wk treatment period.
- Matching Placebo/100 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 100 mg via iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 100 mg dose before considering progression to the 300 mg dose.
- Matching Placebo/300 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 300 mg via iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 300 mg dose before considering progression to the 700 mg dose.
- Matching Placebo/700 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 700 mg via iv infusions separated by 2 wks during the second 24-wk treatment period.
- Total: Total of all reporting groups
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa | Total
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (9.0) | 36.6 (7.0) | 33.7 (8.4) | 37.0 (6.5) | 27.0 (2.2) | 44.0 (8.1) | 36.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 3 | 3 | 0 | 22
  Male | 2 | 5 | 3 | 1 | 1 | 4 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 8 | 11 | 7 | 4 | 4 | 4 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A list of all adverse events is reported in the "Other (Non-Serious) Adverse Events" section. Non-serious AEs were not collected during the Individualized Follow-up Period.
Time Frame: First Treatment Period (FTP): From Visit 3 (Week 0) up to Visit 10 (Week 24); Second Treatment Period (STP): From Visit 10 (Week 24) up to Visit 17 (Week 48); IFUP: up to Visit 26 (Week 104)
Population: Full Analysis Set (FAS): all participants who had been exposed to the investigational product (IP) irrespective of their compliance to the planned course of treatment.
Measure: Number; unit: participants
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
participants
  Weeks 0-24 | 8 | 10 | 7 | 3 | 2 | 2
  Weeks 24-48 | 4 | 5 | 4 | 3 | 4 | 4
  Individualized Follow-up Period | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With the Indicated Critical Adverse Events (CAEs)
Description: A CAE=treatment-related (TR) grade (G) >=3 AE on day of infusion (inf.) preventing inf. to be resumed, a TR G 3 bronchospasm during 1 inf., an AE whose severity becomes G 3 for the third time during 1 inf., infections reported as serious, a TR neurological event consistent with progressive multifocal leukoencephalopathy (PML), any malignancy, and any fatal adverse drug reaction. AE severity (assessed as G 1-5) was classified using the Common Terminology Criteria for Adverse Events v3.0: G 1=mild AE; G 2=moderate AE; G 3=severe AE; G 4=life-threatening or disabling AE; G 5=death related to AE.
Time Frame: FTP: From Visit 3 (Week 0) up to Visit 10 (Week 24); STP: From Visit 10 (Week 24) up to Visit 17 (Week 48); IFUP: up to Visit 26 (Week 104)
Population: FAS
Measure: Number; unit: participants
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
participants
  Week 0-24; Influenza | 0 | 0 | 0 | 1 | 0 | 0
  Week 0-24; Bronchospasm | 0 | 1 | 0 | 0 | 0 | 0
  Week 0-24; Cough | 0 | 1 | 0 | 0 | 0 | 0
  Week 0-24; Rash pruritic | 0 | 1 | 0 | 0 | 0 | 0
  Week 24-48; any CAE | 0 | 0 | 0 | 0 | 0 | 0
  Individualized Follow-up Period; any CAE | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Negative or Unconfirmed Human Anti-human Antibodies (HAHA) in Which Concentrations of Ofa Were Below 500 Nanograms Per Milliliter (ng/ml)
Description: Participants are checked for negative (or a lack of) HAHA at Baseline, and then throughout the study, to ensure that the investigational product is not causing HAHA development. Participants with concentrations of Ofa that are missing or are above 500 nanograms per milliliter (ng/mL) are considered to have unconfirmed HAHA results.
Time Frame: Visit 3 (Week 0), Visit 10 (Week 24), Visit 17 (Week 48) or early withdrawal (EW), and Visit 26 (Week 104)
Population: FAS. Only those participants contributing data at the indicated time points were analyzed (reflected by "n=" in the category titles).
Measure: Number; unit: participants
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
participants
  Week 0; n=8, 8, 2, 4, 3, 4 | 8 | 8 | 2 | 4 | 3 | 4
  Week 24; n=8, 9, 1, 4, 4, 4 | 8 | 9 | 1 | 4 | 4 | 4
  Week 48 or EW, negative; n=8, 11, 7, 4, 3, 4 | 8 | 11 | 7 | 4 | 3 | 1
  Week 48 or EW, unconfirmed, n=8, 11, 7, 4, 3, 4 | 0 | 0 | 0 | 0 | 0 | 3
  IFUP, n=8, 11, 7, 4, 4, 4 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: The investigator performed the physical examination, which included but was not limited to: general appearance and the following body systems: lymph nodes, mouth and throat, lungs, cardiovascular, abdomen, extremities, muscular-skeletal, neurological (apart from multiple sclerosis [a brain and spinal cord disease]), and skin. All abnormal clinically relevant findings such as vein problems (venous varices), disorder of the vertebral column (vertebropathy), increased hearing loss, post operative mark (scar), and chronic skin disorder with no sweat and itching (anhidrotic eczema) were reported.
Time Frame: as for outcome 2
Population: FAS
Measure: Number; unit: participants
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
participants
  Week 0-24; Venous varices on legs | 1 | 0 | 0 | 0 | 0 | 0
  Week 0-24; Vertebropathy | 1 | 0 | 0 | 0 | 0 | 0
  Week 0-24; Obesitas | 1 | 0 | 0 | 0 | 0 | 0
  Week 0-24; Increased hearing loss | 0 | 0 | 1 | 0 | 0 | 0
  Week 0-24; Post operative scar | 0 | 0 | 1 | 0 | 0 | 0
  Week 0-24; Anhidrotic eczema | 0 | 0 | 0 | 0 | 0 | 1
  Week 24-48; Venous varices on legs | 1 | 0 | 0 | 0 | 0 | 0
  Week 24-48; Vertebropathy | 1 | 0 | 0 | 0 | 0 | 0
  Week 24-48; Obesitas | 1 | 0 | 0 | 0 | 0 | 0
  Week 24-48; Acne vulgaris | 0 | 1 | 0 | 0 | 0 | 0
  Week 24-48; Post operative scar | 0 | 0 | 1 | 0 | 0 | 0
  IFUP; Any physical examination finding | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Basophils, Eosinophils, Leukocytes, Monocytes, Lymphocytes, Neutrophils, and Platelet Count at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for hematology assessment. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in basophils, eosinophils, leukocytes, monocytes, lymphocytes, neutrophils, and platelets count was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Week 104 for the IFUP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48); IFUP: Visit 26 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Giga (10^9) per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 7 | 3 | 4 | 4
Giga (10^9) per liter
  Week 0-24, Basophils; n=7, 10, 7, 3, 3, 4 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 0-24, Eosinophils; n=8, 10, 6, 2, 3, 4 | 0 (0.05) | -0.05 (0.13) | 0.02 (0.15) | 0 (0) | -0.23 (0.21) | 0.03 (0.05)
  Week 0-24, Leukocytes; n=8, 10, 7, 3, 4, 4 | 0.7 (1.6) | 0.6 (2.4) | -0.1 (3.3) | -0.3 (1.6) | 0.7 (5.9) | 0.4 (0.7)
  Week 0-24, Lymphocytes; n=8, 10, 7, 3, 3, 4 | 0.15 (1.03) | -0.36 (0.67) | -0.19 (0.78) | -0.37 (0.31) | -0.60 (0.79) | 0.12 (0.21)
  Week 0-24, Monocytes; n=8, 10, 7, 3, 3, 4 | 0.20 (0.31) | -0.07 (0.23) | 0.00 (0.20) | 0.07 (0.06) | -0.40 (0.17) | 0.05 (0.10)
  Week 0-24, Neutrophils; n=8, 10, 7, 3, 3, 4 | 0.4 (0.9) | 1 (2.2) | 0 (3.8) | -0.1 (1.5) | -0.8 (1.7) | 0.2 (0.7)
  Week 0-24, Platelets; n=8, 10, 7, 3, 4, 4 | 0.8 (33.3) | 10.8 (44.0) | 7.6 (39.7) | 0.3 (29.5) | 5.8 (36.2) | -4.8 (34.8)
  Week 24-48, Basophils; n=8, 8, 5, 3, 2, 3 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 24-48, Eosinophils; n=8, 8, 5, 3, 2, 4 | 0 (0.05) | -0.04 (0.16) | 0.04 (0.09) | -0.07 (0.06) | -0.20 (0.28) | 0.03 (0.13)
  Week 24-48, Leukocytes; n=8, 10, 7, 3, 3, 4 | 0.5 (1.1) | -0.1 (1.7) | -0.3 (1.1) | -0.9 (0.6) | -3.7 (1.7) | 0.9 (0.9)
  Week 24-48, Lymphocytes; n=8, 8, 6, 3, 2, 4 | -0.11 (0.36) | -0.28 (0.47) | 0.15 (0.36) | -0.50 (0.20) | -0.65 (0.78) | -0.25 (0.45)
  Week 24-48, Monocytes; n=8, 8, 6, 3, 2, 4 | -0.20 (0.07) | -0.01 (0.12) | 0.02 (0.17) | 0.03 (0.06) | -0.04 (0.28) | 0.13 (0.25)
  Week 24-48, Neutrophils; n=8, 8, 6, 3, 2, 4 | 0.7 (1.2) | 0.2 (1.8) | -0.4 (1.0) | -0.4 (0.4) | -2.9 (1.3) | 1.0 (0.7)
  Week 24-48, Platelets; n=8, 10, 7, 3, 3, 4 | -6.5 (17.3) | -16.3 (74.2) | -10.1 (14.7) | -13.7 (20.6) | -34.3 (47.3) | -11.0 (38.4)
  Week 0-104, Basophils; n=1, 0, 0, 0, 0, 0 | 0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 0-104, Eosinophils; n=1, 0, 0, 0, 0, 0 | 0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 0-104, Leukocytes; n=1, 0, 0, 0, 0, 0 | 1.30 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 0-104, Lymphocytes; n=1, 0, 0, 0, 0, 0 | -0.60 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 0-104, Monocytes; n=1, 0, 0, 0, 0, 0 | 0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 0-104, Neutrophils; n=1, 0, 0, 0, 0, 0 | 1.90 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 0-104, Platelets; n=1, 0, 0, 0, 0, 0 | -20.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

6. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Erythrocyte Count at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for assessment of erythrocyte count. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in erythrocyte count was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48); IFUP: Visit 26 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Pico (10^12) per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 7 | 3 | 4 | 4
Pico (10^12) per liter
  Week 24; n=8, 10, 7, 3, 4, 4 | 0.06 (0.25) | -0.11 (0.33) | -0.02 (0.23) | -0.09 (0.20) | -0.06 (0.42) | 0.07 (0.12)
  Week 48; n=8, 10, 7, 3, 3, 4 | 0.05 (0.26) | 0.12 (0.34) | 0.12 (0.25) | 0.01 (0.43) | 0.06 (0.18) | 0.09 (0.04)
  Week 104; n=1, 0, 0, 0, 0, 0 | -0.08 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

7. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Hematocrit at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for hematocrit assessment. Hematocrit is the percentage of blood volume (BV) that is occupied by red blood cells (RBCs). Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in hematocrit was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline. Hematocrit is measured as a percentage, i.e., volume (V) of red blood cells per volume of blood.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48); IFUP: Visit 26 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of BV occupied by RBCs
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 7 | 3 | 4 | 4
Percentage of BV occupied by RBCs
  Week 24; n=8, 10, 7, 3, 4, 4 | -0.00 (0.03) | 0.01 (0.03) | -0.01 (0.02) | -0.02 (0.02) | 0.02 (0.04) | 0.01 (0.01)
  Week 48; n=8, 10, 7, 3, 3, 4 | 0.01 (0.02) | 0.02 (0.03) | 0.00 (0.03) | 0.01 (0.05) | 0.01 (0.01) | 0.02 (0.01)
  Week 104; n=1, 0, 0, 0, 0, 0 | 0.01 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

8. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Hemoglobin Count at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for assessment of hemoglobin count. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in hemoglobin was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48); IFUP: Visit 26 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles/liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 7 | 3 | 4 | 4
Millimoles/liter
  Week 24; n=8, 10, 7, 3, 4, 4 | 0.1 (0.5) | -0.3 (0.7) | -0.0 (0.5) | -0.4 (0.4) | -0.1 (0.8) | 0.2 (0.2)
  Week 48; n=8, 10, 7, 3, 3, 4 | 0.1 (0.5) | 0.1 (0.7) | 0.2 (0.5) | -0.3 (1.1) | 0.0 (0.3) | 0.5 (0.3)
  Week 104; n=1, 0, 0, 0, 0, 0 | 0.10 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

9. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Albumin at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for assessment of albumin count. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 104 for the IFUP) in albumin was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48); IFUP: VIsit 26 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
grams per liter
  Week 24; n=8, 10, 6, 4, 4, 4 | -0.6 (2.5) | -0.5 (2.5) | 1.3 (1.2) | -1.6 (3.4) | -1.2 (6.1) | 2.0 (2.4)
  Week 48; n=8, 11, 7, 4, 3, 4 | 0.1 (2.5) | -0.2 (3.1) | 1.4 (3.0) | -1.1 (5.7) | 0.4 (4.0) | 1.1 (1.5)
  Week 104; n=1, 0, 0, 0, 0, 0 | -2.00 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

10. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Alkaline Phosphatase, Aspartate Aminotransferase (AST), and Alanine Transaminase (ALT) at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for the assessment of alkaline phosphatase, AST, and ALT. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48); IFUP: up to Visit 26 (Week 104)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
Units per liter
  Week 24, Alkaline phosphatase; n=8, 10, 6, 4, 4, 4 | 4.8 (9.0) | 3.8 (11.9) | 2.7 (8.3) | 13.0 (20.2) | 2.3 (10.6) | 8.8 (8.3)
  Week 24, AST; n=8, 10, 6, 4, 4, 4 | 3.6 (5.1) | 1.6 (6.3) | -0.2 (3.1) | -9.5 (28.6) | 4.3 (3.2) | -1.0 (6.1)
  Week 24, ALT; n=8, 10, 6, 4, 4, 4 | 7.1 (10.2) | 4.7 (10.0) | -1.7 (6.4) | 7.3 (24.4) | 5.3 (5.4) | 0 (13.0)
  Week 48, Alkaline phosphatase; n=8, 11, 7, 4, 3, 4 | 7.6 (10.7) | 3.1 (8.8) | 9.1 (12.6) | 5.3 (17.7) | 5.7 (7.6) | 12.5 (12.9)
  Week 48, AST; n=8, 11, 7, 4, 3, 4 | 0.6 (2.6) | 1.5 (3.0) | 0.3 (2.5) | -13.3 (28.5) | 0.7 (4.7) | 3.3 (10.7)
  Week 48, ALT; n=8, 11, 7, 4, 3, 4 | 2.8 (5.3) | 0.6 (4.7) | 0.6 (7.4) | -4.3 (9.3) | 0.7 (8.1) | 8.0 (20.4)
  Week 104, Alkaline phosphatase; n=1,0,0,0,0,0 | 16.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, AST; n=1, 0, 0, 0, 0, 0 | 2.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, ALT; n=1, 0, 0, 0, 0, 0 | 2.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

11. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Bicarbonate, Glucose, Potassium, Sodium, and Urea at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for the assessment of bicarbonate, glucose, potassium, and urea. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: as for outcome 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimoles per liter
Groups:
- Matching Placebo/300 mg Ofa: Matching placebo was administered as two iv infusions separated by 2 wks during the first 24-wk treatment period. Ofa was administered as two doses of 300 mg via iv infusions separated by 2 wks during the second 24-wk treatment period. An IDMC evaluated the safety data at Week 4 for participants receiving the 300 mg dose before consideAfter completing Week 48 of the second treatment period or withdrawing from the study for any reason, participants entered an Individualized Follow-up Period (IFUP) in which they were monitored for B cell and IgG normalization until individual study termination.ring progression to the 700 mg dose.
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
millimoles per liter
  Week 24, Bicarbonate; n=8, 10, 6, 4, 4, 4 | 0.6 (2.2) | -1.1 (2.6) | -0.6 (2.5) | 1.5 (3.2) | -2.0 (1.3) | -0.6 (4.0)
  Week 24, Glucose; n=8, 10, 7, 4, 4, 4 | -0.12 (0.59) | 0.39 (1.37) | 0.64 (1.23) | 0.21 (0.42) | 0.08 (0.63) | -0.22 (0.50)
  Week 24, Potassium; n=8, 10, 6, 4, 4, 4 | -0.07 (0.35) | 0.06 (0.52) | 0.03 (0.27) | -0.63 (1.01) | -0.20 (0.63) | -0.00 (0.16)
  Week 24, Sodium; n=8, 10, 6, 4, 4, 4 | 0.4 (2.7) | -0.5 (2.8) | -1.2 (1.3) | 0.5 (1.7) | 0.8 (2.1) | 0.5 (2.1)
  Week 24, Urea; n=8, 10, 6, 4, 4, 4 | 0.5 (1.6) | -0.8 (1.6) | 0.4 (1.5) | -0.6 (0.8) | -0.7 (2.1) | -0.1 (0.4)
  Week 48, Bicarbonate; n=8, 11, 7, 4, 4, 4 | -0.0 (2.9) | -0.7 (2.8) | 0.6 (1.3) | 0.6 (0.2) | 1.9 (3.1) | 1.0 (2.3)
  Week 48, Glucose; n=8, 10, 7, 4, 2, 4 | 0.10 (0.50) | 0.25 (0.95) | -0.05 (0.51) | 0.09 (0.56) | -0.64 (0.44) | 0.27 (0.79)
  Week 48, Potassium; n=8, 10, 6, 4, 4, 4 | 4.21 (0.11) | 4.43 (0.44) | 4.18 (0.34) | 4.23 (0.32) | 3.98 (0.10) | 4.20 (0.32)
  Week 48, Sodium; n=8, 11, 7, 4, 3, 4 | -2.3 (1.6) | -0.07 (3.1) | 0.7 (1.0) | -0.5 (3.7) | -0.7 (1.2) | 0.8 (1.0)
  Week 48, Urea; n=8, 11, 7, 4, 3, 4 | 0.13 (1.40) | -0.05 (1.32) | -0.19 (0.68) | -0.30 (1.04) | 1.00 (2.20) | -0.17 (0.46)
  Week 104, Bicarbonate; n=1, 0, 0, 0, 0, 0 | -1.00 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, Glucose; n=1, 0, 0, 0, 0, 0 | 1.77 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, Potassium; n=1, 0, 0, 0, 0, 0 | 0.00 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, Sodium; n=1, 0, 0, 0, 0, 0 | 1.00 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, Urea; n=1, 0, 0, 0, 0, 0 | 1.00 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

12. Primary Outcome: Change From Baseline (Week 0 for the FTP,Week 24 for the STP, and Week 0 for the IFUP) in Bilirubin and Creatinine at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for the assessment of bilirubin and creatinine. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: as for outcome 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
Micromoles per liter (µmol/L)
  Week 24, Bilirubin; n=8, 10, 5, 4, 4, 4 | 0.7 (5.2) | -0.0 (4.0) | 1.2 (2.2) | 0.5 (4.0) | -2.6 (3.5) | 0.3 (5.3)
  Week 24, Creatinine; n=8, 10, 6, 4, 4, 4 | 3.2 (11.8) | -0.1 (7.6) | 2.5 (4.7) | 2.5 (5.7) | -2.9 (7.8) | -1.2 (4.0)
  Week 48, Bilirubin; n=8, 10, 6, 4, 2, 4 | 1.5 (4.9) | -0.1 (4.8) | 1.5 (3.5) | 0.7 (3.4) | -2.8 (1.0) | 0.6 (2.8)
  Week 48, Creatinine; n=8, 11, 7, 4, 3, 4 | 3.0 (8.7) | -1.9 (5.3) | -0.3 (4.1) | 3.5 (6.7) | -5.0 (6.5) | 2.0 (12.5)
  Week 104, Bilirubin; n=1, 0, 0, 0, 0, 0 | -4.70 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, Creatinine; n=1, 0, 0, 0, 0, 0 | 11.5 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

13. Primary Outcome: Change From Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) in Immunoglobins at Week 24 (FTP), Week 48 (STP), and Week 104 (IFUP)
Description: Blood samples of participants were collected for the assessment of antibodies produced by B-cells (immunoglobins): immunoglobulin A, immunoglobin G, and immunoglobin M. Change from Baseline (Week 0 for the FTP, Week 24 for the STP, and Week 0 for the IFUP) was calculated as the value at Visit 10 (Week 24) for the FTP, the value at Visit 17 (Week 48) for the STP, and the value at Visit 26 (Week 104) for the IFUP minus the value at Baseline.
Time Frame: as for outcome 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 7 | 4 | 4 | 4
grams per liter
  Week 24, IGA; n=8, 10, 6, 4, 4, 4 | 0.05 (0.16) | 0.08 (0.16) | 0.40 (0.40) | -0.07 (0.18) | 0 (0.44) | 0.49 (0.35)
  Week 24, IGG; n=8, 10, 6, 4, 4, 4 | -0.6 (1.0) | -0.1 (0.8) | 1.2 (1.0) | -0.5 (1.0) | -0.3 (0.9) | 1.4 (0.9)
  Week 24, IGM; n=8, 10, 6, 4, 4, 4 | -0.09 (0.14) | -0.13 (0.39) | -0.19 (0.09) | 0.25 (0.25) | -0.07 (0.19) | 0.04 (0.08)
  Week 48, IGA; n=8, 11, 7, 4, 3, 4 | 0.08 (0.24) | -0.03 (0.39) | 0.13 (0.11) | -0.00 (0.24) | 0.05 (0.21) | 0.29 (0.26)
  Week 48, IGG; n=8, 11, 7, 4, 3, 4 | -0.8 (1.2) | 0.5 (1.6) | 1.0 (0.7) | -0.6 (1.2) | 0.2 (1.6) | 1.2 (0.6)
  Week 48, IGM; n=8, 11, 7, 4, 3, 4 | -0.17 (0.24) | -0.21 (0.22) | -0.18 (0.24) | -0.24 (0.24) | -0.40 (0.17) | -0.13 (0.04)
  Week 104, IGA; n=1, 0, 0, 0, 0, 0 | -0.23 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, IGG; n=1, 0, 0, 0, 0, 0 | -0.60 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, IGM; n=1, 0, 0, 0, 0, 0 | -0.07 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

14. Primary Outcome: Change From Baseline (Week 0 for the FTP and Week 24 for the STP) in Blood Pressure (BP) at Week 24 (FTP) and Week 48 (STP)
Description: Maximum (systolic) and minimum (diastolic) BP were assessed prior to infusion. Change from Baseline (Week 0 for the FTP and Week 24 for the STP) was calculated as the value at Visit 10 (Week 24) for the FTP and the value at Visit 17 (Week 48) for the STP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
millimeters of mercury
  Week 24, Diastolic BP; n=8, 10, 7, 4, 4, 4 | 5.3 (11.2) | -2.3 (11.1) | -5.4 (9.7) | -3.5 (7.2) | 4.0 (4.9) | -1.8 (2.2)
  Week 24, Systolic BP; n=8, 10, 7, 4, 4, 4 | 11.0 (19.7) | -2.5 (12.3) | -3.1 (14.2) | 1.5 (11.3) | 1.0 (9.0) | -6.5 (9.5)
  Week 48, Diastolic BP; n=8, 11, 7, 4, 3, 4 | 6.6 (4.6) | 2.1 (12.0) | 0.1 (7.8) | 3.0 (4.7) | 3.3 (5.8) | 6.0 (5.8)
  Week 48, Systolic BP; n=8, 11, 7, 4, 3, 4 | 2.0 (14.5) | -2.5 (13.9) | -4.9 (8.2) | -2.3 (7.4) | 1.7 (10.4) | 4.5 (1.0)

15. Primary Outcome: Change From Baseline (Week 0 for the FTP and Week 24 for the STP) in Pulse Rate at Week 24 (FTP) and Week 48 (STP)
Description: The pulse rate of each participant was assessed prior to infusion. Change from Baseline (Week 0 for the FTP and Week 24 for the STP) was calculated as the value at Visit 10 (Week 24) for the FTP and the value at Visit 17 (Week 48) for the STP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
beats per minute
  Week 24; n=8, 10, 7, 4, 4, 4 | -0.3 (11.5) | 1.6 (8.4) | 0.6 (10.7) | 1.3 (13.8) | 2.0 (8.0) | 3.8 (8.1)
  Week 48; n=8, 11, 7, 4, 3, 4 | -0.1 (9.8) | 0.4 (11.9) | -3.0 (10.7) | -5.5 (10.0) | -0.3 (9.5) | 8.0 (5.0)

16. Primary Outcome: Change From Baseline (Week 0 for the FTP and Week 24 for the STP) in Temperature at Week 24 (FTP) and Week 48 (STP)
Description: The temperature of each participant was assessed prior to infusion. Change from Baseline (Week 0 for the FTP and Week 24 for the STP) was calculated as the value at Visit 10 (Week 24) for the FTP and the value at Visit 17 (Week 48) for the STP minus the value at Baseline.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
Degrees Celsius
  Week 24; n=8, 10, 7, 4, 4, 4 | -0.1 (0.5) | 0.1 (0.2) | -0.2 (0.5) | -0.1 (0.4) | 0.3 (0.5) | -0.3 (0.3)
  Week 48; n=8, 11, 7, 4, 3, 4 | -0.1 (0.4) | 0.1 (0.2) | 0.1 (0.5) | -0.1 (0.2) | 0.2 (0.3) | 0.1 (0.3)

17. Primary Outcome: Change From Baseline (Week 0 for the FTP and Week 24 for the STP) in Complement Activation (CH50) at Week 24 (FTP) and Week 48 (STP)
Description: Blood samples of participants were collected for CH50 prior to and 2 hours after dosing, and the samples were sent to a Central Laboratory for analysis: Bio Analytical Research Corporation (BARC). Change from Baseline (Week 0 for the FTP; Week 24 for the STP) was calculated as the value at Weeks 24 (FTP) and 48 (STP) minus the value at Baseline. Ofa depletes (induces the cell death of) B cells. When Ofa binds to a B cell, it induces complement CH50, which in turn causes cell death via cytotoxicity. Therefore, the CH50 levels were measured to ensure that CH50 was being appropriately activated.
Time Frame: FTP: Visit 3 (Week 0) and Visit 10 (Week 24); STP: Visit 10 (Week 24) and Visit 17 (Week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units per milliliter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 7 | 0 | 4 | 2 | 0
Units per milliliter
  Week 24; n=8, 7, 0, 4, 2, 0 | -0.6 (4.1) | -7.1 (12.9) |  | 2.8 (9.1) | -19.5 (24.7) |
  Week 48; n=4, 0, 0, 1, 0, 0 | 3.8 (7.8) | NA (NA) — Data were not collected for this cohort. |  | -31.0 (0) | NA (NA) — Data were not collected for this cohort. |

18. Secondary Outcome: Number of the Indicated Types of Lesions (Ls) Assessed Per Magnetic Resonance Imaging (MRI)
Description: The MRI scan was performed prior to dosing and could be performed up to 4 days prior to Visits 3 and 10. An IDMC reviewed the data. T1 enhancing Ls are enhanced by gadolinium, are considered representative of disease activity/inflammation, and may signify a relapse. Measurement of these Ls is comparative from visit to visit. "Total T1 enhancing Ls" represent the total of the new T1 enhancing Ls over the entire study period. T2 L measurements measure all Ls on the brain in terms of volume and size, measuring for new or enlarging Ls. T1 hypointensive Ls are areas of permanent damage.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
lesions
  Week 24, New (N) T1 enhancing Ls; n=8,11,7,4,4, 4 | 0.13 (0.35) | 0 (0) | 0 (0) | 3.06 (4.66) | 23.50 (43.0) | 2.50 (3.32)
  Week 24, Total T1 enhancing Ls; n=8,11,7,4,4,4 | 0.13 (0.35) | 0.09 (0.30) | 0 (0) | 3.63 (5.02) | 25.75 (46.23) | 4.50 (7.14)
  Week 24, N and/or enlarging T2 Ls; n=8,11,7,4,4,4 | 0.25 (0.71) | 0.09 (0.30) | 0 (0) | 4.00 (6.52) | 25.00 (46.03) | 3.00 (4.24)
  Week 24, N T1 hypointense Ls; n=8,11,7,4, 4,4 | 0 (0) | 0.27 (0.47) | 0.29 (0.49) | 1.50 (3.00) | 5.00 (9.35) | 0.25 (0.50)
  Week 48, N T1 enhancing Ls; n=8,10,7,4,3,4 | 0.13 (0.35) | 0 (0) | 0.29 (0.76) | 0 (0) | 0.33 (0.58) | 0 (0)
  Week 48, Total T1 enhancing Ls; n=8,10,7,4,3,4 | 0.13 (0.35) | 0 (0) | 0.43 (1.13) | 0 (0) | 3.00 (5.20) | 0 (0)
  Week 48, N and/or enlarging T2 Ls; n=8,10,7,4, 3,4 | 0.13 (0.35) | 0 (0) | 0.29 (0.76) | 0 (0) | 0.33 (0.58) | 0 (0)
  Week 48, N T1 hypointense Ls; n=8,10,7,4,3,4 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3.00 (4.36) | 0 (0)
  Week 104, N T1 enhancing Ls; n=1, 0, 0, 0, 0, 0 | 0.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, Total T1 enhancing Ls; n=1, 0, 0, 0, 0,0 | 0.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, N and /or enlarging T2 Ls; n=1,0,0,0,0,0 | 0.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.
  Week 104, N T1 hypointense Ls; n=1, 0, 0, 0, 0, 0 | 0.0 (NA) — Only one participant in this treatment arm was assessed for this parameter at this time point; thus, the standard deviation cannot be calculated. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point. | NA (NA) — No participants were analyzed in this treatment arm at this time point.

19. Secondary Outcome: Total Volume of T2 Lesions at Week 24 and Week 48
Description: The MRI scan should be performed prior to dosing and can be performed up to 4 days prior to Visits 3 and 10. An IDMC reviewed the data. The volume of T2 lesions was not a cumulative volume, but the volume measured at Visit 10 and Visit 17. T2 lesion measurements measure all lesions on the brain in terms of volume and size, measuring for new lesions or enlarging lesions.
Time Frame: Visit 10 (Week 24) and Visit 17 (Week 48)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters cubed
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 11 | 7 | 4 | 4 | 4
millimeters cubed
  Week 24; n=8, 11, 7, 3, 4, 4 | 7898 (8802) | 10323 (8281) | 17399 (11641) | 11290 (11746) | 12194 (18008) | 15039 (8984)
  Week 48; n=8, 10, 7, 4, 3, 4 | 7791 (8878) | 11304 (8269) | 17566 (12413) | 10684 (8903) | 18164 (23696) | 15166 (9060)

20. Secondary Outcome: Ofa Drug Concentration After the First (Visit 3), Second (Visit 4), Third (Visit 10), and Fourth (Visit 11) Intravenous (i.v.) Infusions
Description: The peripheral blood for each participant was collected and analyzed for the concentration of the drug in serum. There were four infusions in the study; the third infusion at Visit 10 represents the first infusion of the second treatment period (Weeks 24-48). Data are presented for the predose concentrations.
Time Frame: Visit 3 (Week 0), Visit 4 (Week 2), Visit 10 (Week 24), and Visit 11 (Week 26). Samples were drawn predose, immediately following the end of infusion, 10 minutes after infusion, 1 hour after infusion, and 2 hours after infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 4 | 4
milligrams per liter
  Week 0; n=8, 10, 6, 0, 0, 0 | 32.3 (9.65) | 85.8 (53.7) | 176 (24.2) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 2; n=8, 10, 6, 0, 0, 0 | 23.4 (19.9) | 64.9 (67.1) | 174 (187) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 24; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 28.9 (8.03) | 43.4 (67.9) | 72.7 (128)
  Week 26; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 21.6 (18.5) | 47.7 (76.9) | 82.4 (144)

21. Secondary Outcome: The Maximum Observed Plasma Concentration (Cmax) After the First (Visit 3), Second (Visit 4), Third (Visit 10), and Fourth (Visit 11) i.v. Infusions
Description: The peripheral blood for each participant was collected and analyzed for Cmax after the first, second, third, and fourth i.v. infusions. Assessment was performed using the noncompartmental method (this analysis is highly dependent on the estimation of total drug exposure).
Time Frame: Visit 3 (Week 0), Visit 4, (Week 2), Visit 10 (Week 24), and Visit 11 (Week 26). Samples were drawn predose, immediately following the end of infusion, 10 minutes after infusion, 1 hour after infusion, and 2 hours after infusion.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 3 | 4
milligrams per liter
  Week 0; n=8, 10, 6, 0, 0, 0 | 36.8 (13.1) | 124 (23.6) | 346 (24.0) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 2; n=8, 10, 6, 0, 0, 0 | 47.7 (14.7) | 157 (25.9) | 452 (28.5) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 24; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 33.2 (13.7) | 137 (40.7) | 312 (24.5)
  Week 26; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 43.5 (25.2) | 210 (54.1) | 416 (24.6)

22. Secondary Outcome: The Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Time Point (AUC(0-t)) After the First (Visit 3), Second (Visit 4), Third (Visit 10), and Fourth (Visit 11) i.v. Infusions
Description: The peripheral blood for each participant was collected and analyzed to estimate the area under the plasma concetration-time curve, AUC(0-t), and was assessed using the non-compartmental method.
Time Frame: Visit 3 (Week 0), Visit 4 (Week 2), Visit 10 (Week 24), and Visit 11 (Week 26). Samples were drawn predose, immediately following the end of infusion, 10 minutes after infusion, 1 hour (hr) after infusion, and 2 hours after infusion.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millgram hour per liter
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 3 | 4
Millgram hour per liter
  Week 0; n=8, 10, 6, 0, 0, 0 | 153 (19.4) | 498 (18.6) | 1528 (20.7) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 2; n=8, 10, 6, 0, 0, 0 | 15559 (34.4) | 63165 (40.6) | 225876 (30.4) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 24; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 123 (8.6) | 624 (32.7) | 1347 (29.1)
  Week 26; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 12763 (29.3) | 71041 (54.9) | 217757 (44.5)

23. Secondary Outcome: Time to Reach Cmax (Tmax) After the First (Visit 3), Second (Visit 4), Third (Visit 10), and Fourth (Visit 11) i.v. Infusions
Description: The peripheral blood for each participant was collected and analyzed for tmax.
Time Frame: Visit 3 (Week 0), Visit 4 (Week 2),Visit 10 (Week 24), and Visit 11 (Week 26). Samples were drawn predose, immediately following the end of infusion, 10 minutes after infusion, 1 hour after infusion, and 2 hours after infusion.
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 3 | 4
hours
  Week 0; n=8, 10, 6, 0, 0, 0 | 5.33 [4.00 to 8.60] | 5.88 [4.17 to 7.67] | 6.00 [5.17 to 9.42] | NA [NA to NA] — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA [NA to NA] — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA [NA to NA] — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 2; n=8, 10, 6, 0, 0, 0 | 4.25 [3.42 to 5.58] | 4.33 [3.52 to 6.13] | 3.83 [3.67 to 4.50] | NA [NA to NA] — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA [NA to NA] — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA [NA to NA] — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Week 24; n=0, 0, 0, 4, 3, 4 | NA [NA to NA] — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA [NA to NA] — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA [NA to NA] — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 4.42 [4.08 to 6.00] | 6.00 [4.17 to 6.92] | 6.54 [4.13 to 8.17]
  Week 26; n=0, 0, 0, 4, 3, 4 | NA [NA to NA] — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA [NA to NA] — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA [NA to NA] — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 3.67 [3.58 to 6.00] | 5.17 [4.08 to 5.50] | 4.50 [3.75 to 5.50]

24. Secondary Outcome: Clearance of Ofa Over the Course of Weeks 0-2 and 24-26
Description: The peripheral blood for each participant was collected and analyzed for clearance. Clearance is the measure of efficiency with which a drug is irreversibly removed form the body. The average clearance over the course of Weeks 0-2 and 24-26 is reported.
Time Frame: Weeks 0-2 and 24-26
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 3 | 4
liters per hour
  Weeks 0-2; n=8, 10, 6, 0, 0, 0 | 0.006 (34.2) | 0.005 (41.0) | 0.003 (30.8) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Weeks 24-26; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 0.008 (29.5) | 0.004 (54.4) | 0.03 (44.4)

25. Secondary Outcome: The Volume of Distribution at Steady State (Vss) of Ofatumumab Over the Course of Weeks 0-2 and 24-26
Description: The peripheral blood for each participant was collected and analyzed for Vss. The average Vss over the course of Weeks 0-2 and 24-26 is reported.
Time Frame: Weeks 0-2 and 24-26
Population: FAS. Only those participants who contributed data at the indicated time points were analyzed (reflected by "n=" in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 3 | 4
liters
  Weeks 0-2; n=8, 10, 6, 0, 0, 0 | 2.48 (20.4) | 2.61 (42.0) | 2.19 (21.3) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Weeks 24-26; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 2.74 (6.54) | 2.20 (68.0) | 2.15 (20.8)

26. Secondary Outcome: Half Life (t1/2) of Ofatumumab in the Terminal Elimination Phase Over the Course of Weeks 0-2 and 24-26
Description: The peripheral blood for each participant was collected and analyzed for half life. Half life is defined as the period of time required for the amount of drug in the body to be reduced by half. The average t1/2 over the course of Weeks 0-2 and 24-26 is reported.
Time Frame: Weeks 0-2 and 24-26
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Number analyzed (Participants) | 8 | 10 | 6 | 4 | 3 | 4
hours
  Weeks 0-2; n=8, 10, 6, 0, 0, 0 | 246 (16.1) | 331 (35.2) | 452 (28.4) | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1. | NA (NA) — Ofa concentrations were only measured in Arms 1-3 during Treatment Period 1. Participants in Arms 4-6 received placebo during Treatment Period 1.
  Weeks 24-26; n=0, 0, 0, 4, 3, 4 | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | NA (NA) — Ofa concentrations were only measured in Arms 4-6 during Treatment Period 2. Participants in Arms 1-3 received placebo during Treatment Period 2. | 241 (23.6) | 342 (16.3) | 453 (49.9)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs are reported for both the first period (FP; Weeks 0-24) and the second period (SP; Weeks 24-48). SAEs were collected during the IFUP (collected/reported up to Week 104); however, non-serious AEs were not.
Description: The duration of B-cell depletion observed following ofatumumab administration makes attribution of an SAE/AE in the SP to placebo versus ofatumumab difficult. Because it may not be appropriate to ascribe events reported in the SP to placebo, SAEs/AEs are reported by treatment sequence rather than by each individual treatment received.
Arm/Group | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo | 300 mg Ofa/Matching Placebo | 700 mg Ofa/Matching Placebo | Matching Placebo/100 mg Ofa | Matching Placebo/300 mg Ofa | Matching Placebo/700 mg Ofa
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/11 | 0/7 | 1/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 8/8 | 10/11 | 7/7 | 3/4 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo (N=8) | 300 mg Ofa/Matching Placebo (N=11) | 700 mg Ofa/Matching Placebo (N=7) | Matching Placebo/100 mg Ofa (N=4) | Matching Placebo/300 mg Ofa (N=4) | Matching Placebo/700 mg Ofa (N=4)
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 Milligrams (mg) Ofatumumab (Ofa)/Matching Placebo (N=8) | 300 mg Ofa/Matching Placebo (N=11) | 700 mg Ofa/Matching Placebo (N=7) | Matching Placebo/100 mg Ofa (N=4) | Matching Placebo/300 mg Ofa (N=4) | Matching Placebo/700 mg Ofa (N=4)
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tonsilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Neck pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
False positive laboratory result (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Hypoaesthesia facial (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Bartholin's cyst removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Antibiotic prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.